CLINICAL TRIAL: NCT01591330
Title: A Particle Size Study of 3 Different Particle Size Test Tablet Formulations Compared to the Reference Tablet Formulation in Healthy Subjects
Brief Title: A Study of LY2140023 in Healthy Males and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12857; H8Y-MC-HBCY (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2012-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pomaglumetad methionil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2140023 Reference Form (Experimental): LY2140023: 80 mg, administered once, orally. There is a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
  Interventions: Drug: LY2140023 Reference form
- LY2140023 Test-Low (Experimental): LY2140023: 80 mg, low particle size, administered once, orally. There is a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
  Interventions: Drug: LY2140023 Test-Low
- LY2140023 Test-Medium (Experimental): LY2140023: 80 mg, medium particle size, administered once, orally. There is a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
  Interventions: Drug: LY2140023 Test-Medium
- LY2140023 Test-High (Experimental): LY2140023: 80 mg, high particle size, administered once, orally. There is a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
  Interventions: Drug: LY2140023 Test-High

INTERVENTIONS:
Drug: LY2140023 Reference form — 80-mg tablet administered orally
  Other Names: LY2140023 Monohydrate (Reference)
  Arms: LY2140023 Reference Form
Drug: LY2140023 Test-Low — 80-mg tablet administered orally
  Other Names: LY2140023 Monohydrate (Test - Low)
  Arms: LY2140023 Test-Low
Drug: LY2140023 Test-Medium — 80-mg tablet administered orally
  Other Names: LY2140023 Monohydrate (Test - Medium)
  Arms: LY2140023 Test-Medium
Drug: LY2140023 Test-High — 80-mg tablet administered orally
  Other Names: LY2140023 Monohydrate (Test - High)
  Arms: LY2140023 Test-High

SUMMARY:
The study will evaluate the effect of different particle size of LY2140023. The study involves 4 single doses of 80 milligrams (mg) LY2140023 taken as 1 tablet by mouth with a washout period of at least 3 days between doses. This study will last approximately 60 days not including screening. Screening is required within 30 days prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* are overtly healthy males or females, as determined by medical history and physical examination
* male participants: agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023 and agree not to donate sperm for 3 months following the last dose of LY2140023
* female participants:

  * female participants of child-bearing potential who test negative for pregnancy at screening and agree to use a reliable method of birth control for the duration of the study and for at least 3 months after the last dose of LY2140023
  * female participants who are of non-childbearing potential (that is, postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy, or confirmed tubal occlusion [not tubal ligation]). Postmenopausal is defined as no menses for at least 1 year, or a plasma follicle stimulating hormone (FSH) value of >40 milli-international units per liter (mIU/mL), unless the participant is taking hormone replacement therapy
* have a body mass index (BMI) of 19 to 32 kilograms per meter squared (kg/m^2), inclusive, at the time of screening
* have clinical laboratory test results within normal reference ranges for the population or investigator site or results with acceptable deviations that are judged to be not clinically significant by the investigator
* have venous access sufficient to allow for blood sampling as per the protocol
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have given written informed consent approved by Lilly and the chosen ethical review board (ERB)

Exclusion Criteria:

* are currently enrolled in or have completed or discontinued within the last 90 days from a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to LY2140023, LY404039, related compounds, or any components of the formulation
* are persons who have previously completed or withdrawn from this study or any other study investigating LY2140023 and have previously received the investigational product
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have an abnormal blood pressure or pulse rate as determined by the investigator
* have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have evidence or any history of significant active neuropsychiatric disease
* have increased risk of seizures based on a history of:

  * one or more seizures (except for a single simple febrile seizure [lacking focality and lasting less than 15 minutes, not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * head trauma with loss of consciousness or a post-concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * uncontrolled migraine or transient ischemic attack (TIA) within 1 year and/or stroke with persistent neurological deficit (focal or diffuse); uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning; TIA is defined as "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * brain surgery
  * electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, or sharp-slow wave complexes, or as locally defined)
  * brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (except hydrocephalus treated by shunt or without neurological deficits).
* show evidence or any history of known substance dependence or abuse at any time (according to Diagnostic and Statistical Manual of Mental Disorders [DSM-IV] diagnosis) or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of human immunodeficiency (HIV) virus infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* intend to use over-the-counter (OTC) or prescription medication within 14 days prior to dosing of LY2140023
* have donated blood of more than 500 milliliters (mL) within the 3 months prior to screening, or plan to donate blood within the 3 months after the last dose
* have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption for 48 hours prior to check-in for each treatment period until discharge in each period (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* have a clinically significant abnormality in the neurological examination
* participants judged prior to randomization to be at suicidal risk by the investigator
* participants who are unwilling to refrain from tobacco- or nicotine-containing products while in the Clinical Research Unit (CRU) or are unable to abide by CRU restrictions
* show evidence of pruritus or skin exfoliation
* have an eosinophil count > 1.5 x 10^9 per liter (L)
* show evidence of active renal disease or creatinine clearance (CrCl) less than 90 milliliters per minute (mL/min) (as calculated by the Cockcroft-Gault equation)
* in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: LY2140023 80 milligrams (mg) reference form (RF) in Period 1, LY2140023 80 mg Test-low in Period 2, LY2140023 80 mg Test-medium in Period 3, LY2140023 80 mg Test-high in Period 4.
  Each LY2140023 dose was administered once, orally. There was a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
- Sequence 2: LY2140023 80 mg Test-low in Period 1, LY2140023 80 mg Test-high in Period 2, LY2140023 80 mg RF Period 3, LY2140023 80 mg Test-medium in Period 4.
  Each LY2140023 dose was administered once, orally. There was a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
- Sequence 3: LY2140023 80 mg Test-high in Period 1, LY2140023 80 mg Test-medium in Period 2, LY2140023 80 mg Test-low in Period 3, LY2140023 80 mg RF in Period 4.
  Each LY2140023 dose was administered once, orally. There was a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
- Sequence 4: LY2140023 80 mg Test-medium in Period 1, LY2140023 80 mg RF in Period 2, LY2140023 80 mg Test-high in Period 3, LY2140023 80 mg Test-low in Period 4.
  Each LY2140023 dose was administered once, orally. There was a minimum 3-day washout period between dosing in one period and dosing in the next dosing period.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 9 | 9 | 9
Received at Least 1 Dose of Study Drug | 8 | 9 | 9 | 9
Completed | 7 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Washout of at Least 3 Days
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 9 | 9 | 9
Completed | 6 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 6 | 9 | 9 | 9
Completed | 5 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Washout of at Least 3 Days
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 5 | 9 | 9 | 9
Completed | 5 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 5 | 9 | 9 | 9
Completed | 5 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout of at Least 3 Days
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 5 | 9 | 9 | 9
Completed | 5 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 5 | 9 | 9 | 9
Completed | 5 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Overall Study: All participants
Arm/Group | Overall Study
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33
  Black or African American | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 71.71 (13.34)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per meter squared (kg/m^2) | 24.73 (3.70)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: All participants who received at least 1 dose of study drug, did not vomit within 5 hours postdose, and have evaluable LY2140023 plasma concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2140023 Reference Form: LY2140023: 80 milligrams (mg), administered once, orally.
- LY2140023 Test-Low: LY2140023: 80 mg, low particle size, administered once, orally.
- LY2140023 Test-Medium: LY2140023: 80 mg, medium particle size, administered once, orally.
- LY2140023 Test-High: LY2140023: 80 mg, high particle size, administered once, orally.
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
nanograms per milliliter (ng/mL) | 277 (25) | 290 (23) | 304 (37) | 284 (29)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Last Time Point of Measurable Concentration (AUC[0-tlast]) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
nanograms*hours per milliliter (ng*h/mL) | 1200 (28) | 1190 (30) | 1210 (32) | 1210 (32)

3. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: All participants who received at least 1 dose of study drug, did not vomit within 5 hours postdose, and have evaluable LY404039 (active moiety) plasma concentration data following administration of LY2140023.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
ng/mL | 476 (14) | 485 (17) | 494 (17) | 490 (16)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Last Time Point of Measurable Concentration (AUC[0-tlast]) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
ng*h/mL | 2640 (17) | 2640 (19) | 2710 (17) | 2700 (16)

5. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (h)
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
hours (h) | 3.00 [2.00 to 5.00] | 3.00 [2.00 to 5.02] | 3.00 [1.00 to 7.00] | 3.00 [2.00 to 5.00]

6. Secondary Outcome: Pharmacokinetics: Terminal Half Life (t1/2) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
h | 2.13 [1.61 to 3.27] | 1.93 [1.55 to 2.95] | 2.02 [1.47 to 3.06] | 2.13 [1.43 to 3.38]

7. Secondary Outcome: Pharmacokinetics: Apparent Total Body Clearance (CL/F) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
liters per hour (L/h) | 66.8 (28) | 67.0 (30) | 65.9 (32) | 66.2 (32)

8. Secondary Outcome: Pharmacokinetics: Volume of Distribution During the Terminal Phase (Vz/F) of LY2140023
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
Liters (L) | 205 (25) | 187 (23) | 192 (26) | 204 (27)

9. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentrations (Tmax) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
h | 4.00 [3.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.00 [1.00 to 6.00] | 4.00 [3.00 to 5.00]

10. Secondary Outcome: Pharmacokinetics: Terminal Half Life (t1/2) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
h | 3.10 [2.46 to 4.24] | 3.05 [2.35 to 4.79] | 2.95 [2.39 to 4.11] | 3.07 [2.71 to 3.85]

11. Secondary Outcome: Pharmacokinetics: Apparent Total Body Clearance (CL/F) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
L/h | 19.3 (17) | 19.3 (19) | 18.9 (17) | 18.9 (16)

12. Secondary Outcome: Pharmacokinetics: Volume of Distribution During the Terminal Phase (Vz/F) of LY404039 (Active Moiety)
Time Frame: Predose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Number analyzed (Participants) | 30 | 28 | 28 | 27
L | 86.3 (28) | 85.0 (32) | 80.4 (26) | 83.6 (23)

ADVERSE EVENTS:
Groups:
- LY2140023 Reference Form: LY2140023: 80 mg, administered once, orally.
Arm/Group | LY2140023 Reference Form | LY2140023 Test-Low | LY2140023 Test-Medium | LY2140023 Test-High
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 17/35 | 15/33 | 12/32 | 16/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2140023 Reference Form (N=35) | LY2140023 Test-Low (N=33) | LY2140023 Test-Medium (N=32) | LY2140023 Test-High (N=32)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (11) | 6 (6) | 7 (7) | 8 (8)
Vomiting (Gastrointestinal disorders) | 5 (8) | 4 (6) | 4 (9) | 6 (10)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 4 (5) | 4 (6) | 5 (8)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days